CLINICAL TRIAL: NCT02635945
Title: A Study to Assess the Efficacy of a 5-day, Once Daily 10- mg PBF-680 Oral Administration Course to Attenuate Allergen Bronchoprovocation-induced Late Asthmatic Responses (LAR) in Asthmatic Patients Controlled on Low-to-medium Dose Inhaled Corticosteroid Maintenance Monotherapy and Inhaled Short Acting Beta-2 Agonist as Rescue Bronchodilator
Brief Title: A Study to Assess the Efficacy of a 5-day, 10- mg PBF-680 Oral Administration on Late Asthmatic Responses (LAR) in Mild to Moderate Asthmatic Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Palobiofarma SL (Industry)
Collaborators: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Hospital de Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IIBSP-PBF-2015-34; 2015-001957-34 (EudraCT Number)
Record Dates: First submitted 2015-10-21; First posted 2015-12-21 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Asthma
Keywords: adenosine A1 receptor antagonist; adenosine receptor modulator; COPD; asthma
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PBF-680 10 mg (Experimental): 2 capsules: PBF-680, 5 mg capsules for oral administration (excipient: 76 mg microcrystalline cellulose).
  Interventions: Drug: PBF-680
- Placebo (Placebo Comparator): 2 capsules: Placebo to PBF-680, as 95.12 mg microcrystalline cellulose capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PBF-680
  Arms: PBF-680 10 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is the second Phase-II trial analyzing efficacy outcomes of PBF-680 in asthmatic subjects, following the supportive data from the proof-of-concept trial on the effect of PBF-680 on airway hyperresponsiveness to adenosine monophasphate (AMP). The purpose of the present study is to provide an assessment on the efficacy of a 5-day treatment course of once daily, orally administered, 10-mg PBF-680 doses, to attenuate "Late Asthmatic Responses" (LAR) as a primary efficacy outcome. The study also aims at analyzing the effect of the PBF-680 treatment course on airway inflammation-related outcomes including airway hyperresponsiveness to AMP at 24 h after allergen bronchoprovocation, plus nitric oxide fraction in exhaled air (FeNO) and airway inflammatory cells counts in induced sputum under the effect of an additional 10-mg PBF-680 dose on the 6th treatment period day. Overall, the study aims at providing evidence on the efficacy of PBF-680 on outcomes, particularly the LAR, that are well established to screen valid drugs for asthma maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults aged ³18, who have signed the informed consent form prior to initiation of any study procedures.
2. Subjects who have controlled asthma, diagnosed and determined as such as per the Global Initiative for Asthma (GINA) guidelines, with low-to-medium dose inhaled corticosteroid (ICS) as maintenance monotherapy and inhaled, short-acting β2-agonist bronchodilator as rescue medication, for a minimum 4-week period before screening visit V1. Controlled asthma under the stated therapy can be the current, stable condition presented at visits V0 and V1 or can be achieved through GINA guideline-based clinical practice through one or more discretionary V0b visits.
3. Subjects must have a body mass index between 18 and 35 kg/m².
4. Subjects must be able to perform acceptable spirometry in accordance with American Thoracic Society (ATS) / European Respiratory Society (ERS) criteria for acceptability and repeatability.

Exclusion Criteria:

1. Current smokers, smokers within six months prior to Visit V1, or subjects with an smoking history greater than 10 packs-years.
2. Asthmatics classed as "intermittent asthma" managed in GINA-1 therapeutic step or asthmatics that need any maintenance controller medication beyond low-to-medium inhaled corticosteroid (ICS).
3. Patients under any immunosuppressive medication whether asthma-related or indicated for any concomitant morbidities.
4. Subjects with a history of life-threatening asthma attacks (i.e. requiring intensive care unit (ICU) admission, orotracheal intubation).
5. Subjects with a history of a respiratory tract infection or an asthma exacerbation requiring the use of antibiotics and/or systemic corticosteroids within 4 weeks prior to visit V1, or who develop a respiratory tract infection or asthma exacerbation during the screening period. In the latter case, the subjects can be re-screened 4 weeks after the last dose of systemic corticosteroid (except for depot corticosteroids; see Table 5.5-1) or antibiotic.
6. Subjects that received bronchial thermoplasty treatment.
7. Subjects with a concomitant pulmonary or thoracic disease other than asthma that may compromise safety or interfere with efficacy outcomes as per site investigator assessment. This includes, but is not limited to, COPD (COPD) attributable to tobacco or α1- antitrypsin deficiency, cystic fibrosis, sarcoidosis, interstitial lung disease, pulmonary hypertension, active pulmonary tuberculosis, or any prior condition that led to pulmonary resection surgery or lung transplantation. Non-cystic fibrosis bronchiectasis without clinically significant morbidity, moderate α1-antitrypsin deficiency without evidence of emphysema or related COPD, or past pulmonary tuberculosis that received proper medical treatment, are acceptable provided that the condition is not expected to interfere with pulmonary function testing as per site investigator assessment.
8. Subjects with any skin condition such as dermographism that may prevent correct interpretation of skin prick allergy tests.
9. Subjects with symptoms of angina pectoris or with a history of confirmed coronary disease or cardiomyopathy.
10. Subjects with A-V block in any degree, sinus bradycardia, tachyarrhythmia, unstable atrial fibrillation, long QT syndrome, corrected QT interval (QTc(F)) interval greater than 450 ms at screening EKG on visit V1, or any other EKG abnormality deemed clinically significant by the investigator.
11. Subjects who have a clinically significant laboratory abnormality at screening blood analysis on visit V2+24h.
12. Subjects with current uncontrolled arterial hypertension.
13. Women of child-bearing potential, unless they are surgically sterile (i.e. bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy), are at least 2 years postmenopausal, practice abstinence, or agree to employ effective contraception from Visit 1 through final visit. Acceptable contraception procedures are oral, transdermal, or implanted contraceptives, intrauterine device, female condom with spermicide, diaphragm with spermicide, or use of a condom with spermicide by the sexual partner.
14. Women supplying lactation.
15. Receipt of any investigational drug or biological therapy within 3 months before randomization in this study, or within 5 half-lives of the investigational agent, whichever is longer. Subjects ever treated with omalizumab or other biological therapies for asthma are not eligible.
16. History of any known immunodeficiency disorder.
17. Subjects with a history of malignancy within the past five years, with the exception of localized basal cell carcinoma of the skin.
18. History of treatment for alcohol or drug abuse within the past year.
19. Subjects with any comorbidity that could affect the safety or efficacy as per site investigator assessment.
20. Subjects not meeting other medication restrictions as stated in Table 5.5-1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Late Asthmatic Response (LAR) , measured as the fall of the forced expiratory volume (FEV1) between 3 and 10 hours postallergen bronchoprovocation | 3-to-10 hour post-allergen bronchoprovocation.

SECONDARY OUTCOMES:
Early Asthmatic Response (EAR), measured as the maximum FEV1 fall from the postdiluent value | within 1 hour post-allergen bronchoprovocation.
hyperresponsiveness to AMP in terms of provocative concentration causing a 20% fall (PC20) increment in response to AMP airway challenge | 24-hour post-allergen bronchoprovocation
Nitric oxide fraction in exhaled air (FeNO) on post-allergen bronchoprovocation day | 6th treatment period day
Total leukocytes per mL in induced sputum on post-allergen bronchoprovocation day | 6th treatment period day
Leukocyte differential counts per mL in induced sputum on post-allergen bronchoprovocation day. | 6th treatment period day
  Leukocyte subpopulations from cytocentrifuged, stained preparations will be counted and expressed as percentage cell numbers per volume unit.
Adverse events | 2 Months
  The occurrence of adverse events will be monitored through the complete study. Adverse events will be recorded with the following information: severity grade (mild, moderate, severe); suspected/unsuspected relationship to the study drug; duration (date and time of onset, defined as precisely as possible, and end date or if continuing at final exam)
Vital signs | 9 times during 2 months
  Vital signs will include radial artery pulse rate (measured for 60 seconds), and systolic and diastolic blood pressure. Pulse rate and blood pressure will be assessed in the right arm after the patient has rested in the sitting position for at least 5 min. Vital sign values will be recorded as notable if: pulse rate <40 or >90 bpm; systolic blood pressure <90 or >140 mmHg; diastolic blood pressure <50 or >90 mmHg.
Number of Participants With Abnormal Laboratory Values | 4 times during 2 months
  On visits V2+24h, V4+24h and V6+24h, venipuncture will be performed for blood laboratory evaluations. The analysis will be performed at the local laboratory, and will include: hemogram with complete blood counts and differential leukocyte counts; clinical biochemistry including electrolytes (sodium, potassium, chloride), glucose, creatinine, urea, aspartate transaminase (AST), alanine transaminase (ALT), gammaglutamyl transpeptidase (GGT) and bilirubin; and serum immunoglobulin E (IgE) (only on visit V2+24h).
Physical examination | 7 times during 2 months
Electrocardiogram (EKG) | 3 times during 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Unitat de Pneumologia Experimental, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No